CLINICAL TRIAL: NCT03619382
Title: An Evaluation Of Healthy Ankle Motion And Morphology In Different Phases Of Simulated Gait Using A Weight-bearing CBCT Scan
Brief Title: An Evaluation Of Healthy Ankle Motion And Morphology
Status: Completed | Type: Observational
Sponsor: Paragon 28 (Industry)
Collaborators: Focus Medical Design and Development (Unknown)
Responsible Party: Sponsor
Other Study IDs: P10-SP-0001
Record Dates: First submitted 2018-07-11; First posted 2018-08-07 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy Ankle
Keywords: ankle
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Subjects identified to have a healthy foot/ankle
  Interventions: Radiation: Cone Beam Computed Tomography; Radiation: Radiographs

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography — Computer tomography (CT) of the foot/ankle for determination of motion and morphology
Radiation: Radiographs — Standard radiographs of the foot/ankle as part of the screening criteria

SUMMARY:
Determine motion and morphology of the healthy ankle during simulated gait.

DETAILED DESCRIPTION:
Healthy volunteers will undergo weight-bearing, cone beam CT scans of their foot/ankle during 3 phases of simulated gait. Motion and morphology of the foot and ankle will be quantified and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. The subject self-reports having a right healthy ankle.
2. The subject agrees to comply with the requirements of the study and complete the study measures.
3. The subject is between the ages of 18 and 65.
4. The subject is willing to provided written informed consent.

Exclusion Criteria:

1. The subject is pregnant.
2. The subject reports having been diagnosed with any form of diabetes.
3. The subject reports having surgery on the right foot, right ankle and/or right knee.
4. The subject reports a history of repeated ankle sprains or injuries to the right ankle.
5. The subject reports a history of instability of the right ankle.
6. The subject reports chronic or recurring pain of the right ankle.
7. The subject is: a prisoner, unable to understand what participation in the study entails, mentally incompetent, and/or known abuser of alcohol and/or drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers who have a healthy ankle
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Relative rotations of bones | 1 day
  Determine relative tri-axial rotations between bones of the foot and ankle using reconstructed 3-dimensional computer models. All rotations will be measured in degrees (°).

SECONDARY OUTCOMES:
Relative translations of bones | 1 day
  Determine relative multi-directional translation between bones of the foot and ankle using reconstructed 3-dimensional computer models. All translations will be measured in mm.
Morphology - size and shape of the bones of the foot and ankle | 1 day
  Evaluate the size and shape of the bones of the foot and ankle using reconstructed 3-dimensional computer models relative to height, weight, body mass index and gender. All distances will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: James Clancy, DPM, Principal Investigator — Orthopedic Center of Palm Beach County
Locations (1):
- Orthopedic Center of Palm Beach County, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Anderle, Mathew R., et al. "A bi-radial approach to define the sagittal geometry of the healthy ankle." Foot and Ankle Surgery (2020). — https://pubmed.ncbi.nlm.nih.gov/33214032/